CLINICAL TRIAL: NCT01351987
Title: An Observational Study of Dutasteride and Alpha-Blocker Combination Therapy in Men With Symptomatic Benign Prostatic Hyperplasia and PSA Level Over 4 ng/mL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Liang-Ming Lee, Superintendent Office, Wanfang Hospital
Other Study IDs: 100006
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
To analyze the change in International Prostate Symptom Score (IPSS) and serum prostate-specific antigen (PSA) level from baseline.

DETAILED DESCRIPTION:
This is a non-interventional, observational and multicenter study. When subjects will be allowed the dutasteride and α-blocker orally once daily for two years by investigator's prescription. They will be invited to this observational study. All eligible subjects can be allowed the prior alpha blockers therapy. Details of acute urinary retention (AUR) and BPH-related prostatic surgery episodes will be recorded at every visit. Subjects will return to the clinic for assessment every 3 months until week 96. The efficacy and safety of combining the 5α-reductase inhibitor (5ARI), dutasteride, and the α-blocker will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Males, age ≧ 50 years
* Clinical diagnosis of BPH by medical history and physical examination, including a digital rectal examination (DRE)
* IPSS score ≧ 8 points and prostate volume ≧ 30 mL
* Total serum PSA ≧ 4.0 ng/mL and ≦ 20 ng/mL at screening
* Previous TRUS-guided biopsy have been done with benign findings and with prostate cancer (CaP) not detected within the past 6 months.
* Dutasteride combination therapy will be allowed by investigator's prescription
* Ability to understand and willingly provide written informed consent

Exclusion Criteria:

* History or evidence of prostate cancer and high grade prostatic intraepithelial neoplasia (HGPIN)
* With symptomatic urinary tract or prostate infection or urinary retention within 3 months prior to entry of study
* Use of finasteride within 6 months of screening visit
* Use of dutasteride within 12 months of screening visit

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Benign Prostatic Hyperplasia male paitents
Sampling Method: Non-Probability Sample
Enrollment: 855 (Estimated)
Dates: Start 2010-12; Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Ming Lee, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan